CLINICAL TRIAL: NCT02905097
Title: Five Year Survival and Functional Assessment of the Triathlon Cementless Total Knee System Using the Tritanium Tibial Baseplate
Brief Title: Post-marketing Surveillance Study of the Triathlon Tritanium Baseplate
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: Stryker GI Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ortho 16-04
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Arthritis
Keywords: Knee arthroplasty, Total; Knee replacement, Total; Survival rate; Osseointegration; Gait
MeSH Terms: conditions — Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroplasty cohort: A cohort of patients who will undergo knee replacement surgery and will receive Triathlon Tritanium (cementless) tibial implant.
  Interventions: Procedure: Knee Replacement

INTERVENTIONS:
Procedure: Knee Replacement — Surgical replacement of arthritic knee with an implant
  Other Names: Knee Arthroplasty

SUMMARY:
The aim of the study is to assess the performance of the cementless Triathlon Tritanium tibial baseplate for total knee replacement, with a minimum follow up of 5 years.

DETAILED DESCRIPTION:
All potential total knee arthroplasty patients from two consultant orthopaedic surgeons at the Golden Jubilee National Hospital (GJNH) will be screened in relation to the inclusion/exclusion criteria. Invitation letters and participant information sheets (PIS) will be sent out to suitable patients who have been referred to the GJNH for total knee replacement (allocated patients) prior to their pre-operative consultation with their surgeon. They will be approached at their consultation visit to seek consent to take part in the study. Patients who have been referred to the GJNH for assessment for a knee replacement (see and treat patients) will be approached only if they are deemed eligible for knee replacement by their consultant, and will be given a copy of the participant information sheet along with the invitation letter. They will be approached for consent to take part in the study at their pre-operative assessment. All patients will be given the opportunity to ask questions about the study before signing the consent form. Consent will be taken by the chief investigator or their delegate, using a signed form.

One hundred patients will be recruited to the study. They will have their surgery performed by one of the participating consultants using the study implant, the Triathlon Tritanium cementless tibial baseplate manufactured by Stryker Corporation.

Participants will receive their standard in-patient care and rehabilitation. Standard hospital care for knee arthroplasty patients is for them to return to the hospital for a post-operative review at 6 weeks and then 1 year and 7 years after operation. Study participants will also be asked to attend the GJNH for two additional research specific appointments at six months and five years. They will be also contacted by post or via telephone to complete a study questionnaire (patient satisfaction) at 3 years post operation.

During the standard care appointments, patients will be reviewed by a member of the arthroplasty team who will collect routine data on the clinical and functional outcomes and implant stability. These data include the Oxford Knee Score (OKS), EURO Quality of life questionnaire (EQ-5D 5L), patient satisfaction and standard radiographic assessment of the implant.

Detailed radiographic analysis will be carried out on radiographs collected as standard and specifically for the study. These will be post-operation at day one (standard), 6 weeks (standard), 6 months (study), 1 year (standard) and the 5 years (study) time points. Study specific radiographic assessment will consist of assessment for radiolucency and osteolysis at specific regions around the tibial and femoral components. Pre-operatively, a standard weight bearing long- leg anterior-posterior (AP) view, lateral view and a skyline view is obtained as per standard care. Post-operatively, standard care consists of a standard weight bearing long-leg AP radiograph at 6 weeks and a short AP and Lateral view at all other reviews.

Study participants will also have two sessions of specialised functional assessment (biomechanical movement analysis and 6-minute walk test) before operation and 1 year after operation during their standard pre and postoperative visits. Biomechanical movement analysis will be carried out in an on-site movement analysis laboratory. Study participants will be required to wear suitable clothing (e.g. tee shirt and shorts) and be barefoot. A number of reflective markers will be attached to specific locations on the body using suitable double sided tape which can be tracked by a number of infrared cameras. participants will be asked to perform the following tasks; walking, stepping up, stepping down, sit-to-stand, stand-to-sit and single leg balance. Each task will be performed at least three times to enable the collection of three good sets of data. In addition, the two stepping tasks will be repeated for each limb. The single leg balance will be performed once for each leg and data will be collected for 30 seconds per limb. A motion capture system will collect limb and torso movements during the task performances while force plates will collect ground reaction forces. The 6-minute walk test requires the participant to walk around a course during a six minute period. They are allowed to have rest breaks for as long and as often as they require. They will be asked to stop walking six minutes after the start of the test and the distance covered during the period will be noted.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral TKA
2. Age 18-75 years
3. BMI <40
4. From one of the following health boards: Ayrshire & Arran, Forth Valley, Greater Glasgow & Clyde, Highland, Lanarkshire or Lothian
5. Suitable to receive the study implant

Exclusion Criteria:

1. Revision of existing knee replacement
2. Previous hip or knee replacement surgery if within the last 12 months
3. Previous ankle surgery
4. Diagnosed osteopenia or osteoporosis
5. Proximal tibial bone defects
6. Unable to give informed consent
7. Unwilling to take part
8. Unable to return to the Golden Jubilee National Hospital for followup appointments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to the Golden Jubilee National Hospital for total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Implant survival at five years | 5 years
  Kaplan-Meier implant survival at 5 years

SECONDARY OUTCOMES:
Component loosening rate | 5 years
  Number of loose components reported
Fracture rate | 5 years
  Number of peri-prosthetic fractures reported
Infection rate | 5 years
  Number of infections reported
Radiolucency | review at 6 weeks, 6 months, 1 and 5 years
  Degree of radiolucent lines around the components
Bone quality | review at 6 weeks, 6 months, 1 and 5 years
  Evidence of bony ingrowth or osteolysis
Component migration | review at 6 weeks, 6 months, 1 and 5 years
  Component movement in mm or degrees from the one day post-operative position
Oxford Knee Score | 6 weeks, 6 months, 1, 3 and 5 years
  Patient-reported knee pain and function
EQ5D-5L | 6 weeks, 6 months, 1, 3 and 5 years
  Patient-reported quality of life
Patient satisfaction | 6 weeks, 6 months, 1, 3, and 5 years
  Patient-reported satisfaction of the knee using a five point Likert scale
Knee function during walking | 1 year
  Knee angles of movement and loads collected using clinical movement analysis
Knee function during stepping up | 1 year
  Knee angles of movement and loads collected using clinical movement analysis
Knee function during stepping down | 1 year
  Knee angles of movement and loads collected using clinical movement analysis
Knee function during sit-to-stand | 1 year
  Knee angles of movement and loads collected using clinical movement analysis
Knee function during stand-sit-to | 1 year
  Knee angles of movement and loads collected using clinical movement analysis
Knee stability during single leg balance | 1 year
  Body sway collected using clinical movement analysis in mm
6 minute walk test | 1 year
  Aerobic endurance assessed by the distance walked (m) in a six minutes
Revision rate | 5 years
  Number of cases revised for any reason or for infection
Surgeon feedback | 1 day post-operatively
  Surgeon assessment of the implant ease of implantation using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ohly, MBBS, FRCSEd, Principal Investigator — nick.ohly@gjnh.scot.nhs.uk
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YH, Park JW, Lim HM, Park ES. Cementless and cemented total knee arthroplasty in patients younger than fifty five years. Which is better? Int Orthop. 2014 Feb;38(2):297-303. doi: 10.1007/s00264-013-2243-4. Epub 2014 Jan 14. PMID 24420155
- [Background] Aprato A, Risitano S, Sabatini L, Giachino M, Agati G, Masse A. Cementless total knee arthroplasty. Ann Transl Med. 2016 Apr;4(7):129. doi: 10.21037/atm.2016.01.34. PMID 27162779
- [Background] Lombardi AV Jr, Berasi CC, Berend KR. Evolution of tibial fixation in total knee arthroplasty. J Arthroplasty. 2007 Jun;22(4 Suppl 1):25-9. doi: 10.1016/j.arth.2007.02.006. PMID 17570273
- [Background] Naudie DD, Ammeen DJ, Engh GA, Rorabeck CH. Wear and osteolysis around total knee arthroplasty. J Am Acad Orthop Surg. 2007 Jan;15(1):53-64. doi: 10.5435/00124635-200701000-00006. PMID 17213382
- [Background] Bassett RW. Results of 1,000 Performance knees: cementless versus cemented fixation. J Arthroplasty. 1998 Jun;13(4):409-13. doi: 10.1016/s0883-5403(98)90006-7. PMID 9645521
- [Background] Albrektsson BE, Carlsson LV, Freeman MA, Herberts P, Ryd L. Proximally cemented versus uncemented Freeman-Samuelson knee arthroplasty. A prospective randomised study. J Bone Joint Surg Br. 1992 Mar;74(2):233-8. doi: 10.1302/0301-620X.74B2.1544959.
- [Background] Berry DJ, Wold LE, Rand JA. Extensive osteolysis around an aseptic, stable, uncemented total knee replacement. Clin Orthop Relat Res. 1993 Aug;(293):204-7. PMID 8339482
- [Background] De Martino I, D'Apolito R, Sculco PK, Poultsides LA, Gasparini G. Total Knee Arthroplasty Using Cementless Porous Tantalum Monoblock Tibial Component: A Minimum 10-Year Follow-Up. J Arthroplasty. 2016 Oct;31(10):2193-8. doi: 10.1016/j.arth.2016.03.057. Epub 2016 Apr 12. PMID 27172865
- [Background] Harwin SF, Kester MA, Malkani AL, Manley MT. Excellent fixation achieved with cementless posteriorly stabilized total knee arthroplasty. J Arthroplasty. 2013 Jan;28(1):7-13. doi: 10.1016/j.arth.2012.06.006. Epub 2012 Jul 31. PMID 22854342
- [Background] Melton JT, Mayahi R, Baxter SE, Facek M, Glezos C. Long-term outcome in an uncemented, hydroxyapatite-coated total knee replacement: a 15- to 18-year survivorship analysis. J Bone Joint Surg Br. 2012 Aug;94(8):1067-70. doi: 10.1302/0301-620X.94B8.28350. PMID 22844047
- [Background] Tai CC, Cross MJ. Five- to 12-year follow-up of a hydroxyapatite-coated, cementless total knee replacement in young, active patients. J Bone Joint Surg Br. 2006 Sep;88(9):1158-63. doi: 10.1302/0301-620X.88B9.17789. PMID 16943464
- [Background] Bagsby DT, Issa K, Smith LS, Elmallah RK, Mast LE, Harwin SF, Mont MA, Bhimani SJ, Malkani AL. Cemented vs Cementless Total Knee Arthroplasty in Morbidly Obese Patients. J Arthroplasty. 2016 Aug;31(8):1727-31. doi: 10.1016/j.arth.2016.01.025. Epub 2016 Jan 29. PMID 26895823
- [Background] Mont MA, Pivec R, Issa K, Kapadia BH, Maheshwari A, Harwin SF. Long-term implant survivorship of cementless total knee arthroplasty: a systematic review of the literature and meta-analysis. J Knee Surg. 2014 Oct;27(5):369-76. doi: 10.1055/s-0033-1361952. Epub 2013 Dec 7. PMID 24318196
- [Background] Fricka KB, Sritulanondha S, McAsey CJ. To Cement or Not? Two-Year Results of a Prospective, Randomized Study Comparing Cemented Vs. Cementless Total Knee Arthroplasty (TKA). J Arthroplasty. 2015 Sep;30(9 Suppl):55-8. doi: 10.1016/j.arth.2015.04.049. Epub 2015 Jun 3. PMID 26118567
- [Background] Khaw FM, Kirk LM, Morris RW, Gregg PJ. A randomised, controlled trial of cemented versus cementless press-fit condylar total knee replacement. Ten-year survival analysis. J Bone Joint Surg Br. 2002 Jul;84(5):658-66. doi: 10.1302/0301-620x.84b5.12692. PMID 12188480
- [Background] Matassi F, Carulli C, Civinini R, Innocenti M. Cemented versus cementless fixation in total knee arthroplasty. Joints. 2014 Jan 8;1(3):121-5. eCollection 2013 Jul-Sep. PMID 25606521
- [Background] Meneghini RM, Mont MA, Backstein DB, Bourne RB, Dennis DA, Scuderi GR. Development of a Modern Knee Society Radiographic Evaluation System and Methodology for Total Knee Arthroplasty. J Arthroplasty. 2015 Dec;30(12):2311-4. doi: 10.1016/j.arth.2015.05.049. Epub 2015 May 29. PMID 26122112
- [Background] Potter GD 3rd, Abdel MP, Lewallen DG, Hanssen AD. Midterm Results of Porous Tantalum Femoral Cones in Revision Total Knee Arthroplasty. J Bone Joint Surg Am. 2016 Aug 3;98(15):1286-91. doi: 10.2106/JBJS.15.00874. PMID 27489319
- [Background] Murray DW, Fitzpatrick R, Rogers K, Pandit H, Beard DJ, Carr AJ, Dawson J. The use of the Oxford hip and knee scores. J Bone Joint Surg Br. 2007 Aug;89(8):1010-4. doi: 10.1302/0301-620X.89B8.19424. PMID 17785736
- [Background] Conner-Spady BL, Marshall DA, Bohm E, Dunbar MJ, Loucks L, Al Khudairy A, Noseworthy TW. Reliability and validity of the EQ-5D-5L compared to the EQ-5D-3L in patients with osteoarthritis referred for hip and knee replacement. Qual Life Res. 2015 Jul;24(7):1775-84. doi: 10.1007/s11136-014-0910-6. Epub 2015 Jan 3. PMID 25555837
- [Background] Ko V, Naylor JM, Harris IA, Crosbie J, Yeo AE. The six-minute walk test is an excellent predictor of functional ambulation after total knee arthroplasty. BMC Musculoskelet Disord. 2013 Apr 24;14:145. doi: 10.1186/1471-2474-14-145. PMID 23617377
- [Background] Jenkins S, Cecins N, Camarri B, Williams C, Thompson P, Eastwood P. Regression equations to predict 6-minute walk distance in middle-aged and elderly adults. Physiother Theory Pract. 2009 Oct;25(7):516-22. doi: 10.3109/09593980802664711. PMID 19925174